CLINICAL TRIAL: NCT06761807
Title: Electrocardiographic and Electrophysiologic Changes After Percutaneous Closure of Atrial Septal Defect
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Fatma Osama Ali Ezz el_deen, Resident doctor, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: EPS and ASD
Record Dates: First submitted 2024-11-19; First posted 2025-01-07 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2025-01

CONDITIONS: ASD; Brady Arrythmia
Keywords: ASD; EPD; Brady arrythmia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Incidence of AV node dysfunction after ASD Closure (Experimental): Determining the incidence of SAN and AVN dysfunction before and after percutaneous ASD closure Comparing ECG and EP parameters of SAN and AVN before and after percutaneous ASD closure
  Interventions: Procedure: Electrophysiology study of heart

INTERVENTIONS:
Procedure: Electrophysiology study of heart — The procedure will be done comparatively for each patient; before the device placement and immediately after the procedure.
  This will be done approaching the same sheath that is placed for ASD device closure (the right femoral vein).
  Only one quadripolar EP catheter will be used, it will be placed in high right atrium then at His bundle.
  The EP study will include:
  Assessment of SAN function using cSNRT (through HRA pacing) Assessment of AH and HV intervals (through His bundle EGM) Assessment of antegrade AVN RP (refractory period) and AVN WP (Wenckebach point) through extra-stimuli and incremental atrial pacing.
  Any inducible arrhythmia will be reported

SUMMARY:
Primary outcomes :

Determining the incidence of SAN and AVN dysfunction before and after percutaneous ASD closure Comparing ECG and EP parameters of SAN and AVN before and after percutaneous ASD closure

Secondary outcomes :

Assessing clinical, echocardiographic and procedural risk factors affecting the AVN function after ASD closure device implantation Determining the incidence of supraventricular arrhythmia inducibility before and after percutaneous ASD closure

DETAILED DESCRIPTION:
Atrial septal defects (ASDs) are one of the most common types of acyanotic congenital heart diseases, comprising 6-10% all congenital heart defects. They represent the most common congenital heart disease diagnosed during adulthood. Secundum ASD is a defect in the fossa ovalis (septum primum), or the superior limb of the septum secundum and is the most common type of ASD (80% of all ASDs).

ASD closure for secundum ASD is recommended regardless of symptoms in patients with evidence of right ventricular (RV) volume overload and no pulmonary arterial hypertension (PAH) or left ventricular (LV) disease. Percutaneous device closure has become the first choice for secundum defect closure in presence of a feasible morphology with a reported low risk of serious complications (≤1% of patients).

Subclinical electrocardiography (ECG) abnormalities, sinoatrial node (SAN) and atrioventricular node (AVN) conduction abnormalities have been reported in patients with ASDs. . The reported incidence of AVN block following ASD device closure varies widely from none up to 6.1%. High-grade AVN block after device closure typically occurs in the first 24-hour post-procedure and may mandates device removal for resolution of heart block.

The mechanism of AVN block after ASD device occlusion could be due to mechanical pressure on the AV node or edema related to trauma. Young age and large defect/device size may be a risk factor for AVN block. Deficient rims of the ASD may also have an impact on development of AVN block.

Whether or not there is a direct impact of ASD device closure on the functional properties of AVN and SAN is not well elucidated. Testing the electrocardiographic and electrophysiologic (EP) parameters of AVN and SAN before and after the procedure could obviously help understanding the real risk

ELIGIBILITY:
Inclusion Criteria:

* All patients presented with secundum ASD eligible for percutaneous transcatheter ASD closure at Assiut university heart hospital

Exclusion Criteria:

* No exclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Estimated)
Dates: Start 2025-01-20 (Estimated); Primary Completion 2026-11-02 (Estimated); Study Completion 2027-11-02 (Estimated)

PRIMARY OUTCOMES:
incidence of SAN dysfunction | baseline
  Determining the incidence of SAN and AVN dysfunction before and after percutaneous ASD closure Comparing ECG and EP parameters of SAN and AVN before and after percutaneous ASD closure
incidence of AVN dysfunction | baseline
  incidence of AVN dysfunction before and after percutaneous ASD closure

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Asakai H, Weskamp S, Eastaugh L, d'Udekem Y, Pflaumer A. Atrioventricular block after ASD closure. Heart Asia. 2016 Aug 1;8(2):26-31. doi: 10.1136/heartasia-2016-010745. eCollection 2016. PMID 27540418
- [Background] Hill SL, Berul CI, Patel HT, Rhodes J, Supran SE, Cao QL, Hijazi ZM. Early ECG abnormalities associated with transcatheter closure of atrial septal defects using the Amplatzer septal occluder. J Interv Card Electrophysiol. 2000 Oct;4(3):469-74. doi: 10.1023/a:1009852312907. PMID 11046184
- [Background] Fischer G, Stieh J, Uebing A, Hoffmann U, Morf G, Kramer HH. Experience with transcatheter closure of secundum atrial septal defects using the Amplatzer septal occluder: a single centre study in 236 consecutive patients. Heart. 2003 Feb;89(2):199-204. doi: 10.1136/heart.89.2.199. PMID 12527678
- [Background] Butera G, Carminati M, Chessa M, Youssef R, Drago M, Giamberti A, Pome G, Bossone E, Frigiola A. Percutaneous versus surgical closure of secundum atrial septal defect: comparison of early results and complications. Am Heart J. 2006 Jan;151(1):228-34. doi: 10.1016/j.ahj.2005.02.051. PMID 16368323
- [Background] Bartakian S, Fagan TE, Schaffer MS, Darst JR. Device closure of secundum atrial septal defects in children <15 kg: complication rates and indications for referral. JACC Cardiovasc Interv. 2012 Nov;5(11):1178-84. doi: 10.1016/j.jcin.2012.07.009. PMID 23174643